CLINICAL TRIAL: NCT05254067
Title: Treatment of Intracranial Wide-neck Aneurysms Using Stent-assisted Coil Embolization with the Codman Enterprise 2 Vascular Reconstruction Device.
Brief Title: Enterprise 2 Vascular Reconstruction Device
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 001.VAS.2017.D
Record Dates: First submitted 2020-11-18; First posted 2022-02-24 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Device recipient
  Interventions: Device: Codman Enterprise 2 Vascular Reconstruction Device

INTERVENTIONS:
Device: Codman Enterprise 2 Vascular Reconstruction Device — a self-expanding nitinol, compliant, closed-cell, recapturable design that can be deployed by a single operator designed to assist in the stent-assisted coil embolization of intracranial aneurysms, specifically those that have a wide neck that would not otherwise maintain the coil embolization material within the aneurysm because of the wide opening at the base of the aneurysm.

SUMMARY:
The primary objective of this study is to collect data regarding the effectiveness of using the Enterprise 2 Reconstruction Device in successfully embolizing intracranial aneurysms with wide neck configuration.

DETAILED DESCRIPTION:
The Codman Enterprise 2 Vascular Reconstruction Device is a self-expanding nitinol, compliant, closed-cell, recapturable design that can be deployed by a single operator. The Codman Enterprise 2 Vascular Reconstruction Device is packaged sterile as a single unit with an introducer sheath and a detachable push wire.

This device was designed to assist in the stent-assisted coil embolization of intracranial aneurysms, specifically those that have a wide neck that would not otherwise maintain the coil embolization material within the aneurysm because of the wide opening at the base of the aneurysm. The Codman Enterprise 2 Vascular Reconstruction Device is approved by the FDA as a Humanitarian Use Device (HUD) in cases of wide-necked saccular cerebral aneurysms.

The primary objective of this study is to collect data regarding the effectiveness of using the Enterprise 2 Reconstruction Device in successfully embolizing intracranial aneurysms with wide neck configuration. Secondly, to determine any safety or delivery problems that may occur, or any adverse patient events that may have previously been undocumented.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years old or older) with intracranial aneurysms with a wide neck (defined as > or = to 4mm, or with a dome to neck ratio of 2:1 or greater).

Exclusion Criteria:

* Small-necked aneurysms, inappropriate for stenting.
* Inability to tolerate anti-platelet medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be initially assessed and if included, will undergo procedure that includes use of the device.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Device Effectiveness-Stent Migration | Patients will be followed for a minimum period of 2 years from the date of the procedure, with planned total duration of 4 years of the study, including follow-up time.
  Prior Observation studies have noted in other stents, that over time, a stent may migrate from its original location, given the flow dynamics and potentially from stent under-sizing. This could potentially disrupt flow through the artery, or even uncover the aneurysm, openining, potentially allowing outflow of embolization coils.
Device Effectiveness- Stent Fore-shortening | Patients will be followed for a minimum period of 2 years from the date of the procedure, with planned total duration of 4 years of the study, including follow-up time.
  If a stent contracts slightly after placement, then it could shorten slightly, particularly if the stent is placed around a tortous corner. In this type of event, generally there is no significant impact to the patient, unless the stent were to shorten and uncover the opening of the aneurysm, potentially allowing embolization coils to come out of the aneurysm.
Device Effectiveness- In-stent stenosis | Patients will be followed for a minimum period of 2 years from the date of the procedure, with planned total duration of 4 years of the study, including follow-up time.
  In this known phenomenon with stents, it is possible that either through local inflammatory reaction or by hyper neointimalization, there can be a buildup of materila on the inner lumen of any stent that is placed.

CONTACTS AND LOCATIONS:
Overall Officials: Bartley Mitchell, MD, Principal Investigator — Methodist Dallas Medical Center Neurovascular Surgery
Locations (1):
- Moody Brain and Spine Institute at Methodist Dallas Medical Center, Dallas, Texas, United States